CLINICAL TRIAL: NCT01963169
Title: Dissemination of a Theory-Based Bone Health Program in Online Communities
Brief Title: Dissemination of a Theory-Based Bone Health Program in Online
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Eun-Shim Nahm, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00041186; R01NR011296 (NIH)
Record Dates: First submitted 2013-04-24; First posted 2013-10-16 (Estimated); Results first posted 2019-12-02 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2019-11

CONDITIONS: Osteoporosis; Health Behaviors
Keywords: Bone Health; Online intervention; Dissemination; Theory-based intervention
MeSH Terms: conditions — Osteoporosis; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TO-BoneHealth Group (Experimental): The group will use the 8-week TO-BoneHealth program, which includes: (1) web learning modules, (2) moderated discussion boards, (3) an Ask-the-Experts section, and (4) a virtual library. In addition, a tool kit and video lecture library are also available to participants. The program will be closed after 8 weeks, and there will be no eNewsletter or bi-weekly follow-ups of bone health behavior goal attainment. After 8 weeks, participants will receive a monthly e-mail informing them of the upcoming surveys.
  Interventions: Behavioral: TO-BoneHealth Program (Bone Power Program)
- TO-BoneHealth Plus Group (Experimental): The group will use the TO-BoneHealth Plus program intervention, which includes the 8-week TO-BoneHealth program followed by bi-weekly theory-based eNewsletters with follow-up of each individual's maintenance of bone health behaviors for 10 months.
  Interventions: Behavioral: TO-BoneHealth Plus Program (Bone Power Plus Program)
- Control Group (No Intervention): No specific intervention will be provided to the control group participants. To keep in contact with participants, a monthly e-mail will be sent to inform them of upcoming follow-up surveys. At the end of the study (upon completion of all five surveys), the control group participants will receive a CD version of the TO-BoneHealth program via mail.

INTERVENTIONS:
Behavioral: TO-BoneHealth Program (Bone Power Program) — The 8-week TO-BoneHealth program include: (1) web learning modules, (2) moderated discussion boards, (3) an Ask-the-Experts section, and (4) a virtual library. In addition, a tool kit and video lecture library are also available to participants. The program will be closed after 8 weeks, and there will be no eNewsletter or bi-weekly follow-ups of bone health behavior goal attainment. After 8 weeks, participants will receive a monthly e-mail informing them of the upcoming surveys.
  Arms: TO-BoneHealth Group
Behavioral: TO-BoneHealth Plus Program (Bone Power Plus Program) — This intervention includes the 8-week TO-BoneHealth program followed by bi-weekly theory-based eNewsletters with follow-up of each individual's maintenance of bone health behaviors for 10 months.
  Arms: TO-BoneHealth Plus Group

SUMMARY:
Bone health is a significant public health issue in the United States. An estimated 10 million Americans age 50 and older are living with osteoporosis, and approximately 50% of women and 25% of men over age 50 will experience an osteoporosis-related fracture in their remaining lifetime. Recent research advancements have produced effective measures to improve and maintain bone health, including exercise, diet, screening tests, pharmacotherapies, and fall prevention strategies. These findings, however, have not been fully incorporated into the daily lives of adults, and many are unaware of the magnitude of bone-health problems. Thus, greater efforts must be made to effectively disseminate evidence-based research findings to improve bone health behaviors of the public. The Internet, with its increasing popularity, can be an effective tool in this endeavor. Despite a great deal of available online health resources, there has been a lack of research investigating effective methods to package and deliver these resources to yield positive public health outcomes. Expanding upon our prior findings and using an innovative approach combining two models of the social cognitive theory (SCT) and the RE-AIM framework (Reach, Effectiveness, Adoption, Implementation, Maintenance), in this proposal, we propose a large scale online study (N = 866) that will compare the long-term impact of two SCT-based online bone health interventions in adults age 50 and older targeting two large online communities. The two interventions are (1) an 8-week SCT-based Online Bone Health (TO-BoneHealth) program and (2) a 12-month TO-BoneHealth Plus program, including the TO-BoneHealth program followed by biweekly theory-based eNewsletters with follow-up of each individual's bone health behaviors ("booster" intervention) for 10 months. The interventions' impact will be assessed on the following the modified RE-AIM framework: (a) Effectiveness (knowledge, selected bone health behaviors, fall incidence, initiation of a discussion about bone health with a primary care provider, eHealth literacy); (b) Reach (number of participants the program reached); (c) Implementation (program usage); and (d) Maintenance (participants' bone health behavior maintenance). With the rapid growth of online communities, findings from this study will significantly contribute to current eHealth practice and research and serve as a dissemination model for other health promotion projects targeting online communities.

DETAILED DESCRIPTION:
Not necessary as the content is covered in other areas of this application.

ELIGIBILITY:
Inclusion Criteria:

* being age 50 or older
* having access to the Internet and e-mail (at home or other places such as public
* libraries, computer lab, etc)
* being able to use the Internet/e-mail independently
* having an e-mail account (or being willing to obtain an e-mail account for this study)
* currently residing in a community setting in the United States
* being able to read and write English

Exclusion Criteria:

* are currently participating in any study(s) on: falls, osteoporosis, and /or nutrition
* had participated in our web-based hip fracture prevention conducted in 2006 - 2007

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 866 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eun-Shim Nahm, PhD, Principal Investigator — University of Maryland, Baltimore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nahm ES, Resnick B, Brown C, Zhu S, Magaziner J, Bellantoni M, Brennan PF, Charters K, Brown J, Rietschel M, An M, Park BK. The Effects of an Online Theory-Based Bone Health Program for Older Adults. J Appl Gerontol. 2017 Sep;36(9):1117-1144. doi: 10.1177/0733464815617284. Epub 2015 Dec 16. PMID 26675352

RESULTS

PARTICIPANT FLOW:
Groups:
- TO-BoneHealth Group: The group will use the 8-week TO-BoneHealth program, which includes: (1) web learning modules, (2) moderated discussion boards, (3) an Ask-the-Experts section, and (4) a virtual library. In addition, a tool kit and video lecture library are also available to participants. The program will be closed after 8 weeks, and there will be no eNewsletter or bi-weekly follow-ups of bone health behavior goal attainment. After 8 weeks, participants will receive a monthly e-mail informing them of the upcoming surveys.
  TO-BoneHealth Program (Bone Power Program): The 8-week TO-BoneHealth program include: (1) web learning modules, (2) moderated discussion boards, (3) an Ask-the-Experts section, and (4) a virtual library. In addition, a tool kit and video lecture library are also available to participants. The program will be closed after 8 weeks, and there will be no eNewsletter or bi-weekly follow-ups of bone health behavior goal attainment.
Period: Overall Study
Arm/Group | TO-BoneHealth Group | TO-BoneHealth Plus Group | Control Group
Started | 301 | 302 | 263
Completed | 242 | 220 | 237
Not Completed | 59 | 82 | 26

BASELINE CHARACTERISTICS:
Population: All participants who were randomized into To-BoneHealth, To-BoneHealth Plus Group and Control groups
Groups:
- Control Group: No specific intervention will be provided to the control group participants.
- Total: Total of all reporting groups
Arm/Group | TO-BoneHealth Group | TO-BoneHealth Plus Group | Control Group | Total
Number analyzed (Participants) | 301 | 302 | 263 | 866
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 213 | 197 | 168 | 578
  >=65 years | 88 | 105 | 95 | 288
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (8.5) | 63 (8.5) | 63.5 (8.5) | 62.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 108 | 91 | 317
  Male | 183 | 194 | 172 | 549
Region of Enrollment [Count of Participants; unit: Participants] — Online data collection
  Participants
    United States | 301 | 302 | 263 | 866

OUTCOME MEASURES:

1. Primary Outcome: Changes in Osteoporosis Knowledge, Self-efficacy/Outcome Expectations for Calcium Intake and Exercise, Health Behaviors (Calcium Intake, Exercise)
Description: The 16-item knowledge on osteoporosis was measured using the revised Osteoporosis Knowledge Test (Range: 0 - 23 [higher better])
  The 11-item self-efficacy for calcium intake subscale of the Osteoporosis Health Belief Scale. (Range: 11 - 110 [higher better])
  The 9-item self-efficacy for Exercise scale. (Range: 0 - 90 [higher better])
  The 6-item calcium intake outcome expectation subscale of the Osteoporosis Health Belief Scale (Range: 6 -30[higher better])
  The 9-item outcome expectations for Exercise Scale. (scoring: range: 9 - 45 [higher better])
Time Frame: 8 weeks
Population: Participants who completed the 8-week survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TO-BoneHealth Group | TO-BoneHealth Plus Group | Control Group
Number analyzed (Participants) | 234 | 226 | 245
units on a scale
  Osteoporosis Knowledge | 19.8 (3.8) | 19.3 (4.1) | 16.7 (4.4)
  CA Intake Self-Efficacy | 89.9 (17.8) | 90.8 (16.1) | 82.7 (21.2)
  CA Intake Outcome Expectations | 23.3 (3.6) | 22.9 (4.0) | 22.5 (3.7)
  Exercise Self-Efficacy | 51.3 (26.4) | 50.8 (25.0) | 47.5 (26.4)
  Exercise Outcome Expectations | 37.8 (7.1) | 37.2 (7.0) | 36.6 (7.6)
Statistical Analysis 1: Comparison: TO-BoneHealth Group vs TO-BoneHealth Plus Group vs Control Group; At 8 week, both intervention groups received the same Bone Power Program intervention. Thus, the analysis for the 8-week outcomes was completed as a two-armed RCT; Test type: Superiority; p < 0.001, Mixed Models Analysis — <0.05 (Threshold); Effect size = 0.54 — The above values are for Knowledge outcome using the revised Osteoporosis Knowledge Test
Statistical Analysis 2: Comparison: TO-BoneHealth Group vs TO-BoneHealth Plus Group vs Control Group; At 8 weeks both intervention groups received the same BonePower intervention. Thus the analysis of 8-week outcome was completed as 2-armed RCT; Test type: Superiority; p < 0.001, Mixed Models Analysis — <0.05 (threshold); Effect size = 0.33 — The above values are for the exercise behavior variable assessed by the 9-item Self-Efficacy for Exercise scale
Statistical Analysis 3: Comparison: TO-BoneHealth Group vs TO-BoneHealth Plus Group vs Control Group; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.009, Mixed Models Analysis — <0.05 (Threshold); Effect size = 0.20 — The above values are for calcium outcome expectation
Statistical Analysis 4: Comparison: TO-BoneHealth Group vs TO-BoneHealth Plus Group vs Control Group; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.002, Mixed Models Analysis — <0.05 (Threshold); Effect Size = 0.18 — The above values are for exercise self-efficacy
Statistical Analysis 5: Comparison: TO-BoneHealth Group vs TO-BoneHealth Plus Group; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.032, Mixed Models Analysis — <0.05 (Threshold); Effect size = 0.14 — The above values are for exercise outcome expectation

2. Primary Outcome: Changes in Calcium Intake
Description: Dietary calcium intake was estimated using a short screening tool developed by Blalock et al. 4. It includes 22 items that assess both frequency and portions various foods that contain calcium and vitamin D. (Higher values are better.)
Time Frame: 8 weeks
Population: Participants who completed the 8-week survey.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | TO-BoneHealth Group | TO-BoneHealth Plus Group | Control Group
Number analyzed (Participants) | 234 | 226 | 245
mg | 1538.4 (1289.2) | 1513.3 (1367.6) | 1278.1 (1059.6)

3. Primary Outcome: Changes in Exercise Time
Description: Exercise behavior was assessed using the 6-item exercise subscale that is part of the Yale Physical Activity Survey. (Higher value is better.)
Time Frame: 8 weeks
Population: Participants who completed the 8-week survey.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | TO-BoneHealth Group | TO-BoneHealth Plus Group | Control Group
Number analyzed (Participants) | 234 | 226 | 245
minutes | 160.6 (196.0) | 137.1 (203.8) | 125.6 (177.9)

ADVERSE EVENTS:
Time Frame: 12 months (throughout the data collection period)
Description: Other Adverse Events: Specific adverse event terms are not collected (Reported as "Not associated/unlikely to be associated to the investigational product/procedure, Unexpected")
Arm/Group | TO-BoneHealth Group | TO-BoneHealth Plus Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/301 | 0/302 | 0/263
Serious Adverse Events (participants affected / at risk) | 0/301 | 0/302 | 0/263
Other Adverse Events (participants affected / at risk) | 14/301 | 25/302 | 7/263
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TO-BoneHealth Group (N=301) | TO-BoneHealth Plus Group (N=302) | Control Group (N=263)
Not associated/unlikely to be associated to the investigational product/procedure, Unexpected (General disorders) | 14 (14) | 25 (25) | 7 (7)

LIMITATIONS AND CAVEATS:
Participants were recruited from two large online communities, and these individuals may have been more familiar with the technology than the general older adult population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No